CLINICAL TRIAL: NCT06527300
Title: A Multicenter, Open-label, Single-arm, Phase II Study of NHWD-870 HCl in Adults and Adolescents with Advanced NUT Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Wenda Pharma Technology LTD. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NHWD-870 HCl-II-02
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor (Phase 1)
Keywords: NHWD-870

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult：NHWD-870 HCl 2mg ； Adolescent：NHWD-870 HCl 1.5mg/2mg (Experimental): Take a fixed dose of NHWD-870 HCl tablets orally.
  Interventions: Drug: NHWD-870 HCl

INTERVENTIONS:
Drug: NHWD-870 HCl — Administered P.O.

SUMMARY:
This is a multicenter, open-label, single-arm, phase II study to evaluate the efficacy, safety, and pharmacokinetics of NHWD-870 HCl in adults and adolescents with advanced NUT cancer.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent signed;
* Subjects must sign and date IEC-approved written informed consent in accordance with the guidelines of the competent authorities and research institutions. Informed consent had to be obtained before any protocol-related procedure that was not part of a participant's routine care was performed.
* Participants must be willing and able to comply with the scheduled visits, treatment protocols, laboratory tests, and other requirements of the study;
* If the subjects were under 18, the participants and their legal guardian authorization signed agreement;
* Both sexes, the first part (adult group) was ≥18 years old and ≤75 years old, the second part (adolescent group) was ≥12 years old and <18 years old;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
* The expected survival period for 3 months or more;
* The histopathological (histopathological diagnosis was the first time according to the tumor tissue pathologic specimens before three years, if more than 3 years should be confirmed in the center of the study to do a biopsy. If, in the investigator's judgment, a biopsy might increase a subject's risk, archival tumor tissue samples up to 3 years old could be collected after discussion with the sponsor) were diagnosed as midline (NUT) cancer by, but not limited to:
* Determination of ectopic NUT protein expression by IHC;
* Detection of NUT gene translocations by fluorescence in situ hybridization (FISH);
* Detection of NUT gene translocations (e.g. BRD3/4 mutation or ≥ 2-fold amplification) by DNA/RNA sequencing.

Exclusion Criteria:

* Prior treatment with a BET inhibitor;
* 3 years before into the group suffering from other malignant tumors, with the exception of removal of cure of basal cell carcinoma, orthotopic bladder cancer or cervical carcinoma in situ;
* The researchers believe the subjects is the need for systemic anti-infection treatment of active infection;
* Patients with clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.
* Imaging shows that the tumor has invaded important blood vessels or the investigators judge that the tumor is likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Completed at least four weeks of treatment, the curative effect evaluation of CR, PR and maintain at least 4 weeks, the proportion of the subjects,up to 5 months;

SECONDARY OUTCOMES:
Duration of response (DoR) | Completed at least four weeks of treatment,first time participants from CR or PR to onset of disease (PD),up to 5 months;
Disease control rate (DCR) | Completed at least four weeks of treatment,tumor curative effect evaluation of CR, PR and SD proportion of subjects,up to 5 months;
Progression-free survival (PFS) | From start studying drug therapy to the disease progression or any reason for the first time the time of death,up to 12 months;
time to remission (TTR) | From the beginning the study drug therapy to ease for the first time (including patients with CR and PR),up to 5 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Three Gorges Hospital Affiliated to Chongqing University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No